CLINICAL TRIAL: NCT03992859
Title: Continuous Serratus Plane Block Added to PECS II vs PECS II Alone for Post Operative Analgesia After Axillary Dissection in Breast Cancer Surgery
Brief Title: Continuous Serrates Plane Block in Axillary Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIMPAX BREAST
Record Dates: First submitted 2018-11-14; First posted 2019-06-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: regional anesthesia
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- serratus catheter (Experimental): Continuous serratus plane block: Ropivacaine 0.2% infusion through a multiple hole catheter (C-Cat Cimpax Denmark)at a fixed dose of 12 ml/h and a multimodal analgesia with acetaminophen and a PCA of morphine
  Interventions: Procedure: Continuous serratus plane block
- standard treatment (No Intervention): Post-operative multimodal analgesia with Acetaminophen and PCA of Morphine

INTERVENTIONS:
Procedure: Continuous serratus plane block — Peripheral nerve catheter placed by the surgeon at the end of surgery
  Arms: serratus catheter

SUMMARY:
Patients undergone to axillary dissection during breast surgery with a PECS I, II block will be randomized to receive either a serratus plane continuous local anesthetic infusion through a multiple hole catheter or nothing. Both groups will receive a patient controlled analgesia with morphine.

DETAILED DESCRIPTION:
84 patients ASA I-III undergoing breast surgery with axillary dissection after modified PECS II block as described by Blanco et al. with Ropivacaine 0.37% 30 ml. General anesthesia with remifentanil 0.1 mcg/Kg/min and Propofol 1.5-2 mg/Kg to facilitate endotracheal intubation will provide for all patients, and maintained with Desflurane and Remifentanil infusion. In case of axillary dissection patient will be randomized to receive either a serratus plane continuous local anesthetic infusion through a multiple hole catheter or nothing. Both groups will receive as intraoperative analgesia 1 g Acetaminophene ev 30 minute before the end of the surgery and 1g. 8h-1 postoperative associated to a patient controlled analgesia with morphine. PCA will set up as follow: bolus 1 mg, lock-out 6 minute, max 20 mg/4h. In the serratus group 10 ml of Ropivacaine 0.5% before fascial closure and a continuous infusion of 12 ml/h of Ropivacaine 0.2% will be provide.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* breast surgery
* informed consent

Exclusion Criteria:

* ASA >3
* allergy to local anesthetic
* opioid administration in the last month
* patient refusal

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 12-48 hours
  A 70% reduction in morphine consumption in the continuous serratus plane block over control

SECONDARY OUTCOMES:
persistent post-surgical pain: numerical rating scale | 3-6 months
  a numerical rating scale (0-10, 0= no pain, 10 = worst imaginable pain),> 4

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Francesco Danelli, MD, Principal Investigator — Azienda USL Reggio Emilia - IRCCS
Locations (1):
- Ausl-Irccs Reggio Emilia, Reggio Emilia, RE, Italy